CLINICAL TRIAL: NCT05029648
Title: Evaluation of Predictive Factors for Psoas Tendinitis After First-line Total Hip Arthroplasty
Acronym: ERATO
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: COS-RGDS-2019-12-054
Record Dates: First submitted 2021-08-16; First posted 2021-08-31 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Psoas Tendinitis
MeSH Terms: interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Simple cohort
  Interventions: Other: Cohort

INTERVENTIONS:
Other: Cohort — Cohort

SUMMARY:
Evaluation of predictive factors for psoas tendinitis after first-line total hip arthroplasty.

A single-centre retrospective study of medical data from the medical records of patients undergoing total hip arthroplasty.

DETAILED DESCRIPTION:
From the medical records of a series of patients operated on for total hip arthroplasty:

Main objective: To assess individual and surgical factors associated with the development of psoas tendinitis.

Secondary objectives:

* To describe the frequency of occurrence of psoas tendinitis
* To describe the outcome of patients who underwent tenotomy.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older, having been informed of the research
* Patient who has had a total hip replacement implanted for at least six months as a first-line treatment
* Patient who has been regularly monitored since the operation and for whom all clinical and radiological data are available during follow-up visits

Exclusion Criteria:

* Patient undergoing revision surgery
* Patient who has indicated his opposition to the use of his medical data
* Patient under legal protection, guardianship or curators

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who have had a total hip replacement for at least six months.
Sampling Method: Non-Probability Sample
Enrollment: 1199 (Actual)
Dates: Start 2011-08-11 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Psoas tendinitis development | 6 months
  Pain remission after tenotomy.

SECONDARY OUTCOMES:
Psoas tendinitis occurrence frequency | 6 months
  Frequency of occurrence of psoas tendinitis
To describe the outcome of patients who have undergone tenotomy | 6 months
  To describe the outcome of patients who have undergone tenotomy

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas BONIN, MD, Principal Investigator — Clinique de la Sauvegarde
Locations (1):
- Clinique de la Sauvegarde, Lyon, France

IPD SHARING:
Plan to Share IPD: No